CLINICAL TRIAL: NCT01568216
Title: "A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of Add-on AMG 747 on Schizophrenia Negative Symptoms"
Brief Title: 20101299: Study to Evaluate the Effect of AMG 747 on Schizophrenia Negative Symptoms
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Toxic Epidermal Necrolysis
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20101299; 2011-004844-23 (EudraCT Number)
Record Dates: First submitted 2012-02-27; First posted 2012-04-02 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Schizophrenia
Keywords: schizophrenia negative symptoms
MeSH Terms: conditions — Schizophrenia | interventions — (R)-2-(4-(phenyl(3-(trifluoromethyl)phenyl)methyl)piperazin-1-yl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AMG 747 - Dose 1 (Experimental)
  Interventions: Drug: AMG 747
- AMG 747 - Dose 2 (Experimental)
  Interventions: Drug: AMG 747
- AMG 747 - Dose 3 (Experimental)
  Interventions: Drug: AMG 747
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 747 — Three dose levels once-daily oral administration
  Arms: AMG 747 - Dose 1; AMG 747 - Dose 2; AMG 747 - Dose 3
Drug: Placebo — Once-daily oral administration
  Arms: Placebo Comparator

SUMMARY:
The purpose of this study is to evaluate the effect of AMG 747 on negative symptoms of schizophrenia in patients who are stable on current antipsychotic treatment. After a run-in period on their current antipsychotic treatment, patients will be randomized to one of the four treatment arms as add-on therapy for a treatment duration of up to 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) schizophrenia
* Total score on the PANSS Marder Negative Symptom Factor Scale (NSFS) ≥20
* Total score on the PANSS Marder Positive Symptom Factor Scale (PSFS) ≤ 30
* Receiving stable antipsychotic therapy for at least 8 weeks prior to screening
* Receiving a stable dose of other psychotropic agents for at least 8 weeks prior to screening
* Subject has had a stable residence or living arrangement for at least 8 weeks prior to screening and the residence or living arrangement is not anticipated to change for the duration of the study
* The subject or subject's legally acceptable representative has provided informed consent.

Exclusion Criteria:

* Current schizoaffective or bipolar disorder, panic disorder, obsessive compulsive disorder, evidence of mental retardation by history or clinical examination or known premorbid IQ ≤ 70
* Clinically significant suicidal ideation or suicide attempts, assaultive behavior or marked changes in mood within the 8 weeks prior to screening, or currently endorsing suicidal ideation in clinical exam
* Substance abuse (with the exception of nicotine or caffeine abuse) within the 8 weeks prior to screening, or during screening
* Substance dependence (with the exception of nicotine or caffeine dependence) within the 6 months prior to screening, or during screening
* Planning to initiate a smoking cessation therapy or otherwise substantially modify nicotine use during the study
* Positive urine drug test for substances of abuse (with the exception of positive screens for prescribed agents such as benzodiazepines).
* Other criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 12 in negative symptoms, as measured by the NSA-16 total score | 12 Weeks
  NSA-16 = 16-item Negative Symptom Assessment Scale, an efficacy scale used for the primary endpoint

SECONDARY OUTCOMES:
Response defined as a ≥ 20% decrease in the NSA-16 total score at week 12 | 12 weeks
  NSA-16 = 16-item Negative Symptom Assessment Scale
Change from baseline to week 12 on the PANSS total score and Marder factor scores | 12 weeks
  Positive and Negative Syndrome Scale (PANSS)
Change from baseline to week 12 on the CGI-S | Week 12
  Clinical Global Impression Severity Scale (CGI-S)
CGI-I scores at week 12 | 12 weeks
  Clinical Global Impression Improvement (CGI-I)
Change on cognition battery | 12 weeks
Change in personal and social functioning | 12 weeks
Change on patient reported outcomes | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (37):
- United States (18):
  - Research Site, Anaheim, California
  - Research Site, Cerritos, California
  - Research Site, Culver City, California
  - Research Site, Garden Grove, California
  - Research Site, Los Angeles, California
  - Research Site, Norwalk, California
  - Research Site, San Bernardino, California
  - Research Site, Torrance, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, North Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Marlton, New Jersey
  - Research Site, Glen Oaks, New York
  - Research Site, Rochester, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Dayton, Ohio
  - Research Site, Houston, Texas
- Australia (3):
  - Research Site, Glenside, South Australia
  - Research Site, Melbourne, Victoria
  - Research Site, Mount Claremont, Western Australia
- Canada (4):
  - Research Site, Calgary, Alberta
  - Research Site, Penticton, British Columbia
  - Research Site, Kingston, Ontario
  - Research Site, Montreal, Quebec
- Research Site, Takapuna, Auckland, New Zealand
- Russia (4):
  - Research Site, Khot'kovo
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Saratov
- Research Site, Singapore, Singapore
- Spain (6):
  - Research Site, Santander, Cantabria
  - Research Site, Barcelona, Catalonia
  - Research Site, Cornellà de Llobregat, Catalonia
  - Research Site, L'Hospitalet de Llobregat, Catalonia
  - Research Site, Madrid, Madrid
  - Research Site, Valencia, Valencia

REFERENCES:
- [Derived] Georgiades A, Davis VG, Atkins AS, Khan A, Walker TW, Loebel A, Haig G, Hilt DC, Dunayevich E, Umbricht D, Sand M, Keefe RSE. Psychometric characteristics of the MATRICS Consensus Cognitive Battery in a large pooled cohort of stable schizophrenia patients. Schizophr Res. 2017 Dec;190:172-179. doi: 10.1016/j.schres.2017.03.040. Epub 2017 Apr 20. PMID 28433500
- [Derived] Dunayevich E, Buchanan RW, Chen CY, Yang J, Nilsen J, Dietrich JM, Sun H, Marder S. Efficacy and safety of the glycine transporter type-1 inhibitor AMG 747 for the treatment of negative symptoms associated with schizophrenia. Schizophr Res. 2017 Apr;182:90-97. doi: 10.1016/j.schres.2016.10.027. Epub 2016 Oct 24. PMID 27789188
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com